CLINICAL TRIAL: NCT07358767
Title: Determining the Impact of Malaria Mass Drug Administration on Malaria Prevalence in Under 15 Children and Pregnant Women
Brief Title: Impact of Malaria Mass Drug Administration on Malaria Prevalence in Under 15 Children and Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NoguchiMIMR 2
Record Dates: First submitted 2026-01-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2021-07

CONDITIONS: Malaria
Keywords: Impact,; malaria; mass drug administration; under 15 children; pregnant women
MeSH Terms: conditions — Malaria; Tooth, Impacted | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: This is a clinical study to be undertaken within a 24-month framework in 8 communities in the Eastern Region of Ghana. The study is designed to compare the baseline to evaluation findings following the interventions. Interventions will be implemented at the community level. An intervention entails testing with RDTs and treatment of all participants with ACTs. 7 interventions and surveys will be undertaken. RDTs are used during interventions to determine the prevalence over time. The study will be conducted in two arms - arm 1 will constitute the MDA intervention arm, while arm 2 will constitute the control arm. there are 4 communities in each arm.
  Arm 1: All participants in the intervention arm are treated with ACTS by CHWs who go from door-to-door during each MDA round.
  Arm 2: in the control arm (no intervention). One rounds of mass screening with RDTs, and treatment of confirmed positive cases with ACTS will be done. (one at baseline and one at evaluation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm: treated Artemeher Lumefantrine (AL) during MDA, Control arm no intervention (Active Comparator): Trained community health workers (CHWs) will conduct door-to-door testing of all participants in intervention arm for malaria parasites using RDTs. This is to determine malaria prevalence. All participants are treated in the intervention arm irrespective of results while only the positive cases will be treated in the control arm. For molecular studies, 200ul (two drops) of blood will be collected on filter paper. Treatment using AL will be conducted following the Ghana National Malaria Treatment Guidelines and followed-up for 4 days (day 1, 2, 3 and 7). Those who receive the treatment will be observed for 30 minutes to ensure that they retain the drug. Those who vomit within this period will have the treatment repeated. Since it is required that patients eat before taking the drug, and household members may not have food when they are tested, some will have to take the medicine later after eating. The research team will pass round to verify that the participants adhering to treatment.
  Interventions: Drug: Artemether-lumefantrine (AL)
- Control arm (No Intervention): There will be intervention in the control arm. CHWs will will conduct two rounds of screening with RDTs at baseline and at evaluation, and treating positive cases with AL. In both arms, if a participant become febrile at any time, they will be tested and treated if confirmed positive for malaria by CHWs or referred to the health facility for further investigation.
  All participants will be tested to determine the prevalence at baseline and endline. This is meant to allow for comparison across sites. Hospital data will also be assessed to determine the impact of the interventions on prevalence of symptomatic malaria parasitaemia in the communities.

INTERVENTIONS:
Drug: Artemether-lumefantrine (AL) — All participants will be treated in the intervention arm irrespective of RDT test results while only the positive cases will be treated in the control arm. For molecular studies, 200ul (two drops) of blood will be collected on filter paper during screening. We will use the Ghana Malaria Treatment Guidelines and followed-up for four days (day 1, 2, 3 and 7). Treated participants will be observed for 30 minutes to ensure that they retain the drug. Those who vomit within this period will repeated treatment. It is required that patients eat before taking the drug, and participants may not have food when they are tested, and would have to take the medicine later after eating. This means that some of the treatment will be unobserved. However, the research team will pass round to vrify participants adherence to treatment. They will ask to see the drug package to ensure that the participants are taking the treatment correctly. This also assures the population that the research team cares.
  Arms: Intervention arm: treated Artemeher Lumefantrine (AL) during MDA, Control arm no intervention

SUMMARY:
This is a clinical trial being done to find better ways to reduce malaria in the community. Malaria is caused by a parasite that is spread by mosquitoes. Some people, especially adults, can carry the malaria parasite without feeling sick, but mosquitoes can still pick up the parasite from them and pass it to others. This makes it hard to stop malaria, particularly among children and pregnant women who are more likely to become ill.

The purpose of this study is to reduce malaria by removing the parasite from as many people in the community as possible, including those who do not have symptoms. By treating everyone, the study aims to reduce the spread of malaria and protect vulnerable groups such as children.

All members of households that agree to take part will be tested for malaria. After testing, everyone will be given malaria medicine, whether or not they feel sick. Participants will be followed up to check for any side effects, such as stomach upset, dizziness, or weakness.

By reducing the amount of malaria parasite in the community, mosquitoes will be less likely to spread malaria from one person to another. If many people participate, malaria illness in the community may decrease, children may stay healthier, and families may spend less money on malaria treatment. The results of this study will help inform future malaria control efforts in similar communities.

DETAILED DESCRIPTION:
Background Rapid scale-up of malaria control interventions in the past decade led to a reasonable decrease in the burden of malaria. The challenges involved with translating research scenarios into implementation are enormous and needs to be clearly understood. In an era with decreasing funding for the health system, it is important to understand not only the economic impact of MDA in the health of under 15 children but also its effect on the partial immunity of the population. Interventions focused on clearing the parasites in asymptomatic individuals in combination with intensive use of other control measures could pave the way for pre-elimination of malaria in endemic communities, especially in an era when the SAR-var-2 virus is ravaging countries across the world. It is important to generate data on the trends on the population acquired anti-malarial immunity over time following MDA. This information could be very important for national malaria control programmes for decision-making and planning scale-up of malaria MDA, either nationally or regionally.

Several studies in Ghana have demonstrated very high levels of asymptomatic malaria in both under five and school age children who have a higher risk of coming down with clinical malaria or continue to serve as a transmission reservoir. IPT of children in a community in the southern parts of the country reportedly reduced the parasite load by 90 % in two years. It has been demonstrated that IPT using SP impacted the production of protective antibodies against malaria. Immuno-suppression has also been reported from experimental studies of artemisinin-derivatives. In Ghana, malaria incidence during the post-intervention period with SP was increased by 62% in infants who received six monthly artesunate + amodiaquine, but this rebound was not seen in children aged one year or more at the time of drug administration. This rebound effect has been observed where the IPT intervention targeted only children leaving out the adults who could be asymptomatic but transmitting. Though this study targets the entire population, the effect of MDA on malaria prevalence will be evaluated in under 15 children. While there are concerns that eliminating the parasite in an endemic community could lead to a rebound or fatalities should the parasites be reintroduced, malaria passive case detection and management will therefore continue to be through the health facilities in the study areas. A recent study in Mali demonstrated that implementing SMC does not affect acquired immunity in children following four rounds.

In a pilot scale-up study of MTTT in the Pakro subdistrict of Ghana, a coverage of more than 79% and a reduction in asymptomatic malaria prevalence of 24% was achieved, and a reduction of 67% in severe anaemia following 3-rounds of MTTT interventions over 1-year only. These results could be further improved if the sub-microscopic parasitaemia is targeted through malaria MDA.

Aims or Objectives of study

Primary objective The main aim of this study is to determine the impact of implementing malaria MDA on malaria prevalence in under 15 children.

Secondary objectives

1. To determine the prevalence of malaria asymptomatic parasitaemia in populations within the Pakro sub district.
2. To assess the effect of malaria MDA on anaemia in under 15 children.
3. To determine the effect of malaria MDA on febrile patients attending health facilities in intervention arm compared to the control arm.
4. To assess the effect of scaling up malaria MDA on malaria antibodies over time in asymptomatic participants.

Study participants:

Community entry activities to sensitise the chiefs and the general population will be conducted at the beginning of the study through meetings and durbars. Once the community leaders and the population have accepted the project, the households will be numbered and participants in each household will be registered during a household census. All households will be given a unique identification code. Everyone within the household will be assigned a code that links them to a particular household and community. After obtaining consent from the household heads, the children will be enrolled but individual assent and consent will be obtained from the other adolescents and adults in the household. The intervention study will target all the household members. The primary outcome will be based on data from all enrolled participants. The effect of the interventions on secondary outcome 1 will be observed in all children aged 2 months to 14 years randomly. In addition, selected under 15 children will have in addition to the other data, their Hb readings taken to assess the level of anaemia. The effect of the interventions on secondary outcome 2 will be observed in all under 15 children. Furthermore, the effect of the intervention on secondary outcomes 3 and 4 will be observed in all participants. The investigators hypothesize that within the study population, the prevalence of asymptomatic parasitaemia should drop by 90% by the end of the first year and by 95% by the end of the second year. This is estimated based on the findings of Ahorlu and colleagues, 2011. In the same light the investigators expect that anaemia should drop by the same proportion.

ELIGIBILITY:
Inclusion Criteria:

* participant must be aged 2 months and above
* be resident in the communities for the period of the study.
* willingness to participate will be proven by a completed and signed consent or assent form.
* Administrative authorization is obtained from the Ghana Health Service and NMIMR IRB.

Exclusion Criteria:

* an individual intends to stay less than one year in the study site or
* an individual who would be absent at some time due to schooling in a boarding school
* has a life-threatening illness (excluding malaria).
* Pregnant women will be tested and if positive referred to the Pokrom Health Centre for appropriate management.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The difference in the prevalence of malaria asymptomatic parasitaemia in children <15 years in the intervention arm compared to the control over time. | From enrolment of participants to end of treatment every two months over 24 months
  The asymptomatic parasitaemia will be compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression).
  Baseline Comparison of Patients: Summary statistics (proportions for categorical variables and means or medians with variances or IQRs for continuous variables) and graphs will be used to detect presence of outliers or unusual observations, and to assess validity of assumptions for statistical tests. Participants will be compared between the two study arms (Intervention communities and control communities) with respect to baseline demographic, clinical and parasitological characteristics. Statistical analysis of the above comparisons for continuous variables will be based on graphs, t-test (or Wilcoxon test), and ANOVA (or Kruskal-Wallis test). Categorical variables will be compared using chi-square tests. All analyses will be performed for the whole population in each arm.

SECONDARY OUTCOMES:
Changes prevalence of anaemia in children <15 years over time | From the enrolment of participants to end of treatment every two months over 24 months
  The difference in prevalence of anaemia in children <15 years in the control arm compared to the control.
  To test for anaemia in children under 15, a portable automated Hemocue photometer will be used to determine the concentration of Haemoglobin. Anaemia in this study is defined as Hb levels less than 10g/dl. Particiapnts with severe anaemia (Hb less than 7g/dl) will be referred to the Health Centre for follow up.
  Comparisons of anaemia in children <15 years across time and study arms will be assessed through Cochrane Armitage test of trends and using chi-square tests (or fisher exact tests) respectively. A binomial logistic regression will be used to test impact of intervention on febrile illnesses.
The difference in symptomatic malaria cases attending health facilities in intervention arm compared to the control arm. | From enrolment of participants to end of treatment every two months over 24 months
  Data for symptomatic parasitaemia at the hospitals and those collected at the community will be compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression). Adjustments for potential confounders including patient's age and use of ITN and baseline temperature will be considered. In addition, these outcomes will also be compared over time using Cochrane Armitage test of trends.
Changes in prevalence of anti-plasmodium antibodies between baseline and evaluation in the intervention and control arm. | From enrolment of participants to end of treatment every two months over 24 months
  Anti PfEMP1 response Total plasma IgG levels were will be measured as to a recently described panel of microsphere bead coupled proteins consisting of 39 P. falciparum derived antigens and tetanus toxoid using the Luminex platform. The panel included VAR2CSA and 35 HIS-tagged CIDR proteins representing all three main groups of PfEMP1. Specifically, 19 different sequence variants of CIDRα1, 12 different variants of CIDRα2-6 and 4 different CIDRδ/γ domain proteins produced in Drosophila Sf9 cells will be included. In addition, the protein array included circumsporozoite protein 1 (CSP1), merozoite surface protein 1 (MSP1) and apical membrane antigen 1 (AMA1). The Luminex-based assays will be performed at NMIMR.

CONTACTS AND LOCATIONS:
Overall Officials: Ndong Ignatius Cheng, PhD, Principal Investigator — NMIMR
Locations (1):
- Pokrom sub district, Koforidua, Eastern Region, Ghana

IPD SHARING:
Plan to Share IPD: No
It is one of the ethical requirements that individual participants' data are kept confidential and therefore cannot be shared.

REFERENCES:
- [Background] Ndong IC, Okyere D, Enos JY, Mensah BA, Nyarko A, Abuaku B, Amambua-Ngwa A, Merle CSC, Koram KA, Ahorlu CS. Prevalence of asymptomatic malaria parasitaemia following mass testing and treatment in Pakro sub-district of Ghana. BMC Public Health. 2019 Dec 3;19(1):1622. doi: 10.1186/s12889-019-7986-4. PMID 31795981
- [Background] Mahamar A, Issiaka D, Youssouf A, Niambele SM, Soumare HM, Attaher O, Barry A, Narum DL, Duffy PE, Greenwood B, Fried M, Dicko A. Effect of 4 years of seasonal malaria chemoprevention on the acquisition of antibodies to Plasmodium falciparum antigens in Ouelessebougou, Mali. Malar J. 2021 Jan 7;20(1):23. doi: 10.1186/s12936-020-03542-9. PMID 33413417
- [Background] Dicko A, Sagara I, Sissoko MS, Guindo O, Diallo AI, Kone M, Toure OB, Sacko M, Doumbo OK. Impact of intermittent preventive treatment with sulphadoxine-pyrimethamine targeting the transmission season on the incidence of clinical malaria in children in Mali. Malar J. 2008 Jul 8;7:123. doi: 10.1186/1475-2875-7-123. PMID 18611271
- [Background] Sarpong N, Owusu-Dabo E, Kreuels B, Fobil JN, Segbaya S, Amoyaw F, Hahn A, Kruppa T, May J. Prevalence of malaria parasitaemia in school children from two districts of Ghana earmarked for indoor residual spraying: a cross-sectional study. Malar J. 2015 Jun 25;14:260. doi: 10.1186/s12936-015-0772-6. PMID 26109461
- [Background] Ndong IC, Okyere D, Enos JY, Amambua-Ngwa A, Merle CSC, Nyarko A, Koram KA, Ahorlu CS. Challenges and perceptions of implementing mass testing, treatment and tracking in malaria control: a qualitative study in Pakro sub-district of Ghana. BMC Public Health. 2019 Jun 6;19(1):695. doi: 10.1186/s12889-019-7037-1. PMID 31170964
- [Background] Boulanger D, Sarr JB, Fillol F, Sokhna C, Cisse B, Schacht AM, Trape JF, Riveau G, Simondon F, Greenwood B, Remoue F. Immunological consequences of intermittent preventive treatment against malaria in Senegalese preschool children. Malar J. 2010 Dec 17;9:363. doi: 10.1186/1475-2875-9-363. PMID 21167018
- [Background] Diawara F, Steinhardt LC, Mahamar A, Traore T, Kone DT, Diawara H, Kamate B, Kone D, Diallo M, Sadou A, Mihigo J, Sagara I, Djimde AA, Eckert E, Dicko A. Measuring the impact of seasonal malaria chemoprevention as part of routine malaria control in Kita, Mali. Malar J. 2017 Aug 10;16(1):325. doi: 10.1186/s12936-017-1974-x. PMID 28797263
- [Background] Organization, W.H., World malaria report 2018. 2018. World Health Organization: Geneva.
- [Background] Organization, W.H., World malaria report 2019
- [Background] Newell K, Kiggundu V, Ouma J, Baghendage E, Kiwanuka N, Gray R, Serwadda D, Hobbs CV, Healy SA, Quinn TC, Reynolds SJ. Longitudinal household surveillance for malaria in Rakai, Uganda. Malar J. 2016 Feb 9;15:77. doi: 10.1186/s12936-016-1128-6. PMID 26861943
- [Background] Bousema T, Okell L, Felger I, Drakeley C. Asymptomatic malaria infections: detectability, transmissibility and public health relevance. Nat Rev Microbiol. 2014 Dec;12(12):833-40. doi: 10.1038/nrmicro3364. Epub 2014 Oct 20. PMID 25329408
- [Background] Lindblade KA, Steinhardt L, Samuels A, Kachur SP, Slutsker L. The silent threat: asymptomatic parasitemia and malaria transmission. Expert Rev Anti Infect Ther. 2013 Jun;11(6):623-39. doi: 10.1586/eri.13.45. PMID 23750733
- [Background] Samuels AM, Awino N, Odongo W, Abong'o B, Gimnig J, Otieno K, Shi YP, Were V, Allen DR, Were F, Sang T, Obor D, Williamson J, Hamel MJ, Patrick Kachur S, Slutsker L, Lindblade KA, Kariuki S, Desai M. Community-based intermittent mass testing and treatment for malaria in an area of high transmission intensity, western Kenya: study design and methodology for a cluster randomized controlled trial. Malar J. 2017 Jun 7;16(1):240. doi: 10.1186/s12936-017-1883-z. PMID 28592250
- [Background] Ahorlu CK, Koram KA, Seakey AK, Weiss MG. Effectiveness of combined intermittent preventive treatment for children and timely home treatment for malaria control. Malar J. 2009 Dec 11;8:292. doi: 10.1186/1475-2875-8-292. PMID 20003357
- [Background] Rao VB, Schellenberg D, Ghani AC. Overcoming health systems barriers to successful malaria treatment. Trends Parasitol. 2013 Apr;29(4):164-80. doi: 10.1016/j.pt.2013.01.005. Epub 2013 Feb 14. PMID 23415933
- [Background] Otupiri, E., D. Yar, and J. Hindin, Prevalence of Parasitaemia, Anaemia and treatment outcomes of Malaria among School Children in a Rural Community in Ghana. Journal of Science and Technology (Ghana), 2012. 32(1): p. 1-10.